CLINICAL TRIAL: NCT03976362
Title: A Phase 3 Study of Pembrolizumab in Combination With Carboplatin/Taxane (Paclitaxel or Nab-paclitaxel) Followed by Pembrolizumab With or Without Maintenance Olaparib in the First-line Treatment of Metastatic Squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Pembrolizumab (MK-3475) With or Without Maintenance Olaparib in First-line Metastatic Squamous Non-small Cell Lung Cancer (NSCLC, MK-7339-008/KEYLYNK-008)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7339-008; MK-7339-008 (Other: MSD Protocol Number); KEYLYNK-008 (Other: MSD); 194894 (Registry Identifier: JAPIC-CTI); 2023-508449-41-00 (Registry Identifier: EU CT); U1111-1298-1950 (Registry Identifier: UTN); 2018-004721-88 (EudraCT Number)
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Squamous Cell, Non-small-cell Lung
Keywords: PD-1; PD L1; PD L2
MeSH Terms: conditions — Carcinoma | interventions — pembrolizumab; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; olaparib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Carboplatin + Taxane + Olaparib (Experimental): For the Induction Phase, participants receive 4 cycles:
  Pembrolizumab 200 mg, intravenous (IV) on Day 1 of each 21-day cycle PLUS carboplatin PLUS a taxane (either paclitaxel or nab-paclitaxel) for 4 cycles (21-day cycles). If the participant has a complete or partial response or stable disease to induction therapy, the participant is randomized to maintenance therapy.
  For the Maintenance Phase, participants receive pembrolizumab IV on Day 1 of each 21-day for up to 31 cycles PLUS maintenance oral olaparib 300 mg twice daily. In the Maintenance Phase, the participant continues to receive maintenance olaparib until centrally verified progressive disease, physician decision or intolerable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Olaparib
- Pembrolizumab + Carboplatin + Taxane + Olaparib Placebo (Active Comparator): For the Induction Phase, participants receive 4 cycles:
  Pembrolizumab 200 mg, intravenous (IV) on Day 1 of each 21-day cycle PLUS carboplatin PLUS a taxane (either paclitaxel or nab-paclitaxel) for 4 cycles (21-day cycles). If the participant has a complete or partial response or stable disease to induction therapy, the participant is randomized to maintenance therapy.
  For the Maintenance Phase, participants receive pembrolizumab IV on Day 1 of each 21-day for up to 31 cycles PLUS matching maintenance olaparib placebo twice daily. In the Maintenance Phase, the participant continues to receive maintenance olaparib placebo until centrally verified progressive disease, physician decision or intolerable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®; ONXAL™
Drug: Nab-paclitaxel — IV infusion
  Other Names: ABRAXANE®
Drug: Olaparib — Tablets
  Other Names: LYNPARZA®
  Arms: Pembrolizumab + Carboplatin + Taxane + Olaparib
Drug: Placebo — Placebo to olaparib, tablets
  Arms: Pembrolizumab + Carboplatin + Taxane + Olaparib Placebo

SUMMARY:
The current study will compare pembrolizumab (MK-3475) plus maintenance olaparib, vs. pembrolizumab plus maintenance olaparib placebo for the treatment of squamous NSCLC. The study's 2 primary hypotheses are:

1. Pembrolizumab plus maintenance olaparib is superior to pembrolizumab plus maintenance olaparib placebo with respect to progression-free survival (PFS) per RECIST 1.1 by blinded independent clinical review (BICR).
2. Pembrolizumab plus maintenance olaparib is superior to pembrolizumab plus maintenance olaparib placebo with respect to overall survival (OS).

As of Amendment 07, there will be no further analyses for OS and patient-reported outcome assessments.

DETAILED DESCRIPTION:
This study has 2 phases: an Induction Phase (4 Cycles) and a Maintenance Phase (Up to 31 cycles of pembrolizumab). In the Induction Phase, participants receive pembrolizumab plus carboplatin plus a taxane (paclitaxel or nab-paclitaxel). In the Maintenance Phase, participants with a partial or complete disease response or with stable disease after completing four cycles of induction therapy and who meet eligibility criteria will be randomly assigned to receive pembrolizumab plus maintenance olaparib OR pembrolizumab plus maintenance olaparib placebo. In the Maintenance Phase, participants randomly assigned to receive pembrolizumab for up to 31 cycles plus maintenance olaparib OR maintenance olaparib placebo until centrally verified progressive disease (PD), intolerable toxicities, or physician decision.

As of Amendment 07, participants actively taking placebo will discontinue taking the placebo intervention and continue in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis squamous NSCLC.
2. Have Stage IV squamous NSCLC.
3. Have measurable disease based on RECIST 1.1.
4. Have not received prior systemic treatment for their advanced/metastatic NSCLC.
5. Have provided archival tumor tissue sample or newly obtained core or incisional biopsy of a tumor lesion not previously irradiated.

   Note: Adequacy of biopsy specimen for the above analyses must be confirmed by the central laboratory before the participant can receive study intervention(s). Submission of another tumor specimen may be required prior to enrolling the participant, if adequate tumor tissue was not provided the first time.
6. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status assessed within 7 days prior to the administration of study intervention
7. Have a life expectancy of at least 3 months.
8. Has adequate organ function.
9. Male and female participants who are not pregnant and of childbearing potential must follow contraceptive guidance during the treatment period and for 180 days afterwards.
10. Male participants must refrain from donating sperm during the treatment period and for 180 days afterwards.

Exclusion Criteria:

1. Has non-squamous histology NSCLC.
2. Has a known additional malignancy that is progressing or has progressed within the past 3 years requiring active treatment.
3. Has known active central nervous system metastases and/or carcinomatous meningitis.
4. Has a known hypersensitivity to any components or excipients of carboplatin, paclitaxel or nab-paclitaxel, or olaparib.
5. Has a severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
6. Has an active autoimmune disease that has required systemic treatment in past 2 years.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy.
8. Has a known history of human immunodeficiency virus (HIV) infection, a known history of hepatitis B infection, or known active hepatitis C virus infection.
9. Has interstitial lung disease, or history of pneumonitis requiring systemic steroids for treatment.
10. Has received prior therapy with olaparib or with any other polyadenosine 5' diphosphoribose (polyADP ribose) polymerization (PARP) inhibitor.
11. Has received prior therapy with an agent directed to programmed cell death ligand 1 (PD-L1), anti PD-L2, or directed to a stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137).
12. Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2026-01-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (178):
- United States (18):
  - Alabama Oncology Bruno Cancer Center ( Site 0001), Birmingham, Alabama
  - Disney Family Cancer Center ( Site 0005), Burbank, California
  - Boca Raton Regional Hospital ( Site 0018), Boca Raton, Florida
  - Mid-Florida Cancer Centers ( Site 0022), Orange City, Florida
  - H. Lee Moffitt Cancer Center and Research Institute ( Site 0024), Tampa, Florida
  - Columbus Regional Research Institute ( Site 0099), Columbus, Georgia
  - Mount Sinai Hospital Medical Center ( Site 0035), Chicago, Illinois
  - Oncology of Northshore ( Site 0036), Rolling Meadows, Illinois
  - Methodists Hospitals/Premier Oncology Hematology Associates ( Site 0039), Merrillville, Indiana
  - MedStar Franklin Square Medical Center ( Site 0044), Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute ( Site 0046), Detroit, Michigan
  - Hattiesburg Clinic ( Site 0051), Hattiesburg, Mississippi
  - Frontier Oncology ( Site 0052), Billings, Montana
  - Bozeman Health Deaconness Cancer Center ( Site 0053), Bozeman, Montana
  - Waverly Hematology Oncology ( Site 0054), Cary, North Carolina
  - Thompson Cancer Survival Center ( Site 2812), Knoxville, Tennessee
  - Renovatio Clinical ( Site 0074), The Woodlands, Texas
  - Cancer Care Northwest ( Site 0083), Spokane Valley, Washington
- Argentina (10):
  - Hospital Italiano Regional del Sur ( Site 0509), Bahía Blanca, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0516), Mar del Plata, Buenos Aires
  - Hospital Britanico de Buenos Aires ( Site 0500), Buenos Aires, Buenos Aires F.D.
  - Instituto Medico Rio Cuarto ( Site 0501), Río Cuarto, Córdoba Province
  - Sanatorio Parque ( Site 0515), Rosario, Santa Fe Province
  - Centro Oncológico de Rosario ( Site 0507), Rosario, Santa Fe Province
  - Centro Medico San Roque ( Site 0506), San Miguel de Tucumán, Tucumán Province
  - Hospital Italiano de Buenos Aires ( Site 0511), Buenos Aires
  - Clínica Universitaria Reina Fabiola ( Site 0505), Córdoba
  - Sanatorio Privado San Geronimo S.R.L ( Site 0510), Santa Fe
- Australia (4):
  - Liverpool Hospital ( Site 1201), Liverpool, New South Wales
  - Southern Medical Day Care Centre ( Site 1200), Wollongong, New South Wales
  - Townsville General Hospital ( Site 1202), Townsville, Queensland
  - Monash Cancer Centre ( Site 1205), Clayton, Victoria
- Austria (5):
  - Innsbruck LKH ( Site 1302), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 1307), Linz, Upper Austria
  - Klinikum Wels-Grieskirchen ( Site 1304), Wels, Upper Austria
  - Social Medical Center - Otto Wagner Hospital ( Site 1301), Vienna, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf ( Site 1300), Vienna
- Brazil (11):
  - Instituto do Cancer do Ceara ( Site 0251), Fortaleza, Ceará
  - Hospital Sao Rafael ( Site 0258), Salvador - BA, Estado de Bahia
  - Oncologica do Brasil ( Site 0256), Belém, Pará
  - Hospital Tacchini ( Site 0265), Bento Gonçalves, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre ( Site 0255), Porto Alegre, Rio Grande do Sul
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 0252), Itajaí, Santa Catarina
  - Hospital de Base de Sao Jose de Rio Preto ( Site 0254), Sao Jose Rio Preto, São Paulo
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0253), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0250), São Paulo
  - Hospital Paulistano - Amil Clinical Research ( Site 0263), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 0260), São Paulo
- Canada (8):
  - Nova Scotia Health Authority ( Site 0103), Halifax, Nova Scotia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0107), Hamilton, Ontario
  - Kingston Health Sciences Centre ( Site 0102), Kingston, Ontario
  - Stronach Regional Cancer Centre ( Site 0100), Newmarket, Ontario
  - CISSS de la Monteregie-Centre ( Site 0101), Greenfield Park, Quebec
  - Hopital Cite de la Sante de Laval ( Site 0105), Laval, Quebec
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0110), Montreal, Quebec
  - CIUSSS de la Mauricie et du Centre du Quebec ( Site 0106), Trois-Rivières, Quebec
- France (9):
  - Centre Hospitalier De Chauny ( Site 1411), Chauny, Aisne
  - CHU Caen ( Site 1406), Caen, Calvados
  - CHU Angers ( Site 1405), Angers, Maine-et-Loire
  - Institut De Cancerologie De Lorraine ( Site 1409), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hopital Robert Schuman ( Site 1402), Vantoux, Moselle
  - Centre Jean Perrin ( Site 1407), Clermont-Ferrand, Puy-de-Dome
  - Centre Hospitalier de Pau ( Site 1412), Pau, Pyrenees-Atlantiques
  - CHU de Rouen ( Site 1403), Rouen, Seine-Maritime
  - Hopital d'Instruction des Armees Begin ( Site 1413), Saint-Mandé, Val-de-Marne
- Germany (13):
  - Studienzentrum Aschaffenburg ( Site 1575), Aschaffenburg, Bavaria
  - Klinikum der LMU ( Site 1550), Munich, Bavaria
  - Klinikum Bogenhausen Staedt. Klinikum Muenchen GmbH ( Site 1573), Munich, Bavaria
  - Universitaetsklinikum Regensburg ( Site 1562), Regensburg, Bavaria
  - Klinikum Wuerzburg Mitte gGmbH ( Site 1559), Würzburg, Bavaria
  - Universitaetsklinikum Frankfurt ( Site 1563), Frankfurt am Main, Hesse
  - Pneumologische Lehrklinik Universitaet Goettingen ( Site 1551), Immenhausen, Hesse
  - Universitaetsmedizin Goettingen ( Site 1557), Göttingen, Lower Saxony
  - Universitaetsklinikum Bonn ( Site 1574), Bonn, North Rhine-Westphalia
  - Kliniken Essen Mitte ( Site 1567), Essen, North Rhine-Westphalia
  - InVo-Institut fuer Versorgungsforschung in der Onkologie ( Site 1564), Koblenz, Rhineland-Palatinate
  - Helios Klinikum Erfurt GmbH ( Site 1552), Erfurt, Thuringia
  - Katholisches Marienkrankenhaus gGmbH ( Site 1572), Hamburg
- Japan (15):
  - National Hospital Organization Nagoya Medical Center ( Site 0806), Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital ( Site 0803), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0801), Kashiwa, Chiba
  - Kurume University Hospital ( Site 0814), Kurume, Fukuoka
  - Kanazawa University Hospital ( Site 0811), Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center ( Site 0807), Yokohama, Kanagawa
  - Sendai Kousei Hospital ( Site 0812), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 0804), Hirakata, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 0813), Sakai, Osaka
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0802), Sunto-gun, Shizuoka
  - National Hospital Organization Kyushu Medical Center ( Site 0805), Fukuoka
  - Niigata Cancer Center Hospital ( Site 0808), Niigata
  - Okayama University Hospital ( Site 0810), Okayama
  - Osaka International Cancer Institute ( Site 0809), Osaka
  - The Cancer Institute Hospital of JFCR ( Site 0800), Tokyo
- Mexico (6):
  - Investigacion Onco Farmaceutica S de RL de CV ( Site 0300), La Paz, Baja California Sur
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0334), Guadalajara, Jalisco
  - Arke Estudios Clinicos ( Site 0333), Mexico City, Mexico City
  - Axis Heilsa S. de R.L. de C.V. ( Site 0301), Monterrey, Nuevo León
  - CLIMERS Clinical Medical Research ( Site 0306), Orizaba, Veracruz
  - FAICIC Clinical Research ( Site 0303), Veracruz
- New Zealand (2):
  - MidCentral DHB Palmerston North Hospital ( Site 1102), Palmerston North, Manawatu-Wanganui
  - Capital & Coast District Health Board - Wellington Hospital ( Site 1101), Wellington
- Poland (7):
  - Przychodnia Lekarska Komed ( Site 2416), Konin, Greater Poland Voivodeship
  - MED-POLONIA Sp. z o.o. ( Site 2419), Poznan, Greater Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im Jana Pawla II ( Site 2420), Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc ( Site 2417), Olsztyn, Lower Silesian Voivodeship
  - Wielospecjalistyczny Szpital SPZOZ w Zgorzelcu ( Site 2404), Zgorzelec, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Szpital Rejonowy im. dr Jozefa Rostka ( Site 2402), Racibórz, Silesian Voivodeship
- Romania (6):
  - Cardiomed SRL Cluj-Napoca ( Site 2504), Cluj-Napoca, Cluj
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 2507), Cluj-Napoca, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 2508), Craiova, Dolj
  - Policlinica Oncomed SRL ( Site 2505), Timișoara, Timiș County
  - S.C.Focus Lab Plus S.R.L ( Site 2502), Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf Apostol Andrei ( Site 2501), Constanța
- Russia (13):
  - Russian Oncological Research Center n.a. N.N.Blokhin of MoH ( Site 2000), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 2024), Moscow, Moscow
  - Moscow Research Oncology Institute named after P.A. Hertsen ( Site 2009), Moscow, Moscow
  - FSAI Treatment and Rehabilitation Centre of the MoH and SD of RF ( Site 2006), Moscow, Moscow
  - Moscow Regional Oncological Dispensary ( Site 2028), Balashikha, Moscow Oblast
  - Nizhniy Novgorod Region Oncology Dispensary ( Site 2026), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Budgetary Healthcare Institution of Omsk Region Clinical Oncology Dispensary-Chemotherapy #1 ( Site, Omsk, Omsk Oblast
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 2016), Samara, Samara Oblast
  - SBHI Leningrad Regional Clinical Hospital ( Site 2002), Saint Petersburg, Sankt-Peterburg
  - SPb Central Clinical Railway Hospital ( Site 2003), Saint Petersburg, Sankt-Peterburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 2004), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City Clinical Oncological Dispensary ( Site 2001), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 2021), Kazan', Tatarstan, Respublika
- South Korea (9):
  - National Cancer Center ( Site 1006), Goyang-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 1003), Gyeonggi-do, Kyonggi-do
  - Ajou University Hospital ( Site 1004), Suwon, Kyonggi-do
  - Gyeongsang National University Hospital ( Site 1005), Jinju, Kyongsangnam-do
  - Chungbuk National University Hospital ( Site 1002), Cheongju-si, North Chungcheong
  - Asan Medical Center ( Site 1007), Songpa-gu, Seoul
  - Seoul National University Hospital ( Site 1000), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1001), Seoul
  - Korea University Guro Hospital ( Site 1008), Seoul
- Spain (6):
  - Hospital Duran i Reynals ( Site 1710), L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario de Jaen ( Site 1713), Jaén, La Coruna
  - Hospital Sant Creu i Sant Pau ( Site 1711), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 1716), Madrid
  - Complejo Hospitalario de Malaga ( Site 1714), Málaga
  - Hospital Universitario Virgen Macarena ( Site 1712), Seville
- Taiwan (6):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 0907), Kaohsiung City
  - China Medical University Hospital ( Site 0904), Taichung
  - National Cheng Kung University Hospital ( Site 0905), Tainan
  - National Taiwan University Hospital ( Site 0900), Taipei
  - Mackay Memorial Hospital ( Site 0902), Taipei
  - Chang Gung Medical Foundation.Linkou Branch ( Site 0903), Taoyuan District
- Turkey (Türkiye) (9):
  - Namik Kemal Universitesi Tip Fakultesi ( Site 2100), Tekirdağ, Tekirdas
  - Baskent Unv. Adana Uyg. ve Arast. Hastanesi ( Site 2101), Adana
  - Gazi Universitesi Tip Fakultesi ( Site 2104), Ankara
  - Ankara Sehir Hastanesi ( Site 2105), Ankara
  - Bezmialem Vakif Univ. Tıp Fakultesi Hastanesi Tibbi Onkoloji Bolumu ( Site 2107), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 2103), Istanbul
  - Ege Universitesi Tip Fakultesi ( Site 2109), Izmir
  - Erciyes Universitesi Tip Fakultesi ( Site 2108), Kayseri
  - Ondokuz Mays Üniversitesi Tp Fakültesi Hastanesi-Oncology ( Site 2106), Samsun
- Ukraine (12):
  - Cherkasy Regional Oncology Dispensary ( Site 2225), Cherkasy, Cherkasy Oblast
  - City Clinical Hosp.4 of DCC ( Site 2215), Dnipro, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 2218), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 2226), Kharkiv, Kharkivs’ka Oblast’
  - Regional Centre of Oncology-Thoracic organs ( Site 2219), Kharkiv, Kharkivs’ka Oblast’
  - PP PPC Acinus Medical and Diagnostic Centre ( Site 2223), Kropyvnytskyi, Kirovohrad Oblast
  - Medical Center Asklepion LLC ( Site 2243), Khodosovka, Kyivska Oblast
  - Kyiv City Clinical Oncology Centre ( Site 2224), Kyiv, Kyivska Oblast
  - Medical and Diagnostic Centre LLC Dobryi Prognoz ( Site 2227), Kyiv, Kyivska Oblast
  - MI Odessa Regional Oncological Centre ( Site 2222), Odesa, Odesa Oblast
  - Central City Clinical Hospital ( Site 2221), Uzhhorod, Zakarpattia Oblast
  - Medical Center Verum ( Site 2228), Kyiv
- United Kingdom (9):
  - Southend University Hospital NHS Foundation Trust ( Site 1913), Westcliff-on-Sea, Essex
  - Barts Health NHS Trust - St Bartholomew s Hospital ( Site 1923), London, London, City of
  - Chelsea and Westminster Hospital ( Site 1901), London, London, City of
  - Newcastle Freeman Hospital ( Site 1902), Newcastle upon Tyne, Newcastle Upon Tyne
  - West Suffolk Hospitals NHS Trust ( Site 1919), Bury St Edmunds, Suffolk
  - Western General Hospital, Edinburgh ( Site 1924), Edinburgh, United Kingdom
  - Singleton Hospital ( Site 1909), Swansea, Wales
  - Colchester General Hospital ( Site 1911), Colchester, Worcestershire
  - Birmingham Heartlands Hospital ( Site 1910), Birmingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Hochmair M, Schenker M, Cobo Dols M, Kim TM, Ozyilkan O, Smagina M, Leonova V, Kato T, Fedenko A, De Angelis F, Rittmeyer A, Gray JE, Greystoke A, Aggarwal H, Huang Q, Zhao B, Lara-Guerra H, Nadal E. Pembrolizumab With or Without Maintenance Olaparib for Metastatic Squamous NSCLC That Responded to First-Line Pembrolizumab Plus Chemotherapy. J Thorac Oncol. 2025 Feb;20(2):203-218. doi: 10.1016/j.jtho.2024.10.012. Epub 2024 Oct 28. PMID 39477187
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26267&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of an Induction, Maintenance and Posttreatment phase. For induction, eligible participants were enrolled to receive pembrolizumab and carboplatin plus paclitaxel or nab-paclitaxel. Participants who met additional criteria were randomized 1:1 into a maintenance phase to receive either pembrolizumab combined with olaparib or pembrolizumab combined with placebo. In the posttreatment phase, participants were either followed up or administered a second course of pembrolizumab.
Groups:
- Pembrolizumab (Pembro) + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase): Participants received Pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) on Day 1 of each 21-day cycle for 4 cycles PLUS Carboplatin Area Under Curve (AUC) 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles PLUS investigator's choice of either Paclitaxel (200 mg/m^2 Q3W on Day 1 of each 21-day cycle for 4 cycles or Nab-paclitaxel (100 mg/m^2 Q3W on Days 1, 8, 15 of each 21-day cycle for 4 cycles). Participants may then randomize to one of the blinded treatment arms.
- Pembro + Olaparib (Maintenance Phase): This arm includes participants who randomized following completion of the induction period. After the induction period, participants received pembrolizumab IV on Day 1 of each 21-day for up to 31 cycles PLUS maintenance oral olaparib 300 mg twice daily. In the Maintenance Phase, the participant continued to receive maintenance olaparib until centrally verified progressive disease, physician decision or intolerable toxicity.
  Participants treated with pembrolizumab who completed 35 cycles of pembrolizumab during the study with stable disease (SD), complete response (CR), or partial response (PR), and without a current adverse event (AE), may have been eligible for retreatment with up to an additional 17 cycles (approximately 1 year) of pembrolizumab if they experienced radiographic disease progression after stopping treatment in the Maintenance Phase.
- Pembro + Placebo (Maintenance Phase): This arm includes participants who randomized following completion of the induction period. After the induction period, participants received pembrolizumab IV on Day 1 of each 21-day for up to 31 cycles PLUS matching maintenance olaparib placebo twice daily. In the Maintenance Phase, the participant continued to receive maintenance olaparib placebo until centrally verified progressive disease, physician decision or intolerable toxicity.
  Participants treated with pembrolizumab who completed 35 cycles of pembrolizumab during the study with SD, CR, or PR, and without a current AE, may have been eligible for retreatment with up to an additional 17 cycles (approximately 1 year) of pembrolizumab if they experienced radiographic disease progression after stopping treatment in the Maintenance Phase.
Period: Induction Phase
Arm/Group | Pembrolizumab (Pembro) + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase) | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Started | 851 | 0 | 0
Completed | 591 | 0 | 0
Not Completed | 260 | 0 | 0
Not completed — Failure to Meet Maintenance Randomization Criteria | 198 | 0 | 0
Not completed — Death | 62 | 0 | 0
Period: Maintenance Phase
Arm/Group | Pembrolizumab (Pembro) + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase) | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Started | 0 | 296 (Per protocol, eligible participants were randomized to one of the maintenance treatment arms. Not all participants from the induction period continued into the randomized maintenance phase.) | 295 (Per protocol, eligible participants were randomized to one of the maintenance treatment arms. Not all participants from the induction period continued into the randomized maintenance phase.)
Pembro + Olaparib/Placebo (Second Course Pembro Only) | 0 | 7 | 9
Completed | 0 | 0 | 0
Not Completed | 0 | 296 | 295
Not completed — Participants Ongoing | 0 | 106 | 103
Not completed — Withdrawal by Subject | 0 | 4 | 4
Not completed — Failure To Meet Randomization Criteria | 0 | 0 | 1
Not completed — Death | 0 | 186 | 187

BASELINE CHARACTERISTICS:
Population: Pembro + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase): All enrolled participants who were not randomized into maintenance phase Pembro + Olaparib (Maintenance Phase): Intention-to-Treat (ITT) Population which included all randomized participants post induction phase Pembro + Placebo (Maintenance Phase): Intention-to-Treat (ITT) Population which included all randomized participants post induction phase
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab (Pembro) + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase) | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase) | Total
Number analyzed (Participants) | 260 | 296 | 295 | 851
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (8.6) | 64.2 (8.8) | 64.6 (7.8) | 64.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 60 | 170
  Male | 205 | 241 | 235 | 681
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 47 | 48 | 129
  Not Hispanic or Latino | 211 | 239 | 235 | 685
  Unknown or Not Reported | 15 | 10 | 12 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 9 | 11 | 25
  Asian | 76 | 63 | 51 | 190
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 4 | 4 | 3 | 11
  White | 164 | 214 | 219 | 597
  More than one race | 2 | 1 | 3 | 6
  Unknown or Not Reported | 9 | 5 | 7 | 21
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all selfcare but unable to carry out any work activities, up & about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled, cannot carry on any selfcare, totally confined to bed or chair or Grade 5: Dead. Population: Data for this baseline measure were not collected for the induction phase per protocol.
  Participants
    Grade 0: number analyzed (Participants) | 0 | 296 | 295 | 591
    Grade 0 | 0 | 83 | 82 | 165
    Grade 1: number analyzed (Participants) | 0 | 296 | 295 | 591
    Grade 1 | 0 | 213 | 213 | 426
Response [Count of Participants; unit: Participants] — Participants last scan before randomization assessed based on blinded independent central review (BICR) Assessment per (Response Evaluation Criteria in Solid Tumors RECIST) 1.1 of the latest evaluable scan obtained prior to randomization. Population: Data for this baseline measure were not collected for the induction phase per protocol.
  Participants
    Complete Response (CR)l/Partial Response (PR): number analyzed (Participants) | 0 | 296 | 295 | 591
    Complete Response (CR)l/Partial Response (PR) | 0 | 211 | 218 | 429
    Stable Disease (SD): number analyzed (Participants) | 0 | 296 | 295 | 591
    Stable Disease (SD) | 0 | 84 | 76 | 160
    Progressive Disease (PD): number analyzed (Participants) | 0 | 296 | 295 | 591
    Progressive Disease (PD) | 0 | 1 | 0 | 1
    Missing: number analyzed (Participants) | 0 | 296 | 295 | 591
    Missing | 0 | 0 | 1 | 1
Programmed Cell Death-Ligand 1 (PD-L1) Expression Level: Tumor Proportion Score (TPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Participants with a TPS ≥50% were classified as PD-L1 strongly positive and participants with a TPS <50% were classified as not strongly positive.
  Participants
    Tumor Proportion Score (TPS)<50% | 187 | 208 | 208 | 603
    TPS≥50% | 64 | 85 | 85 | 234
    Not Evaluable | 5 | 2 | 2 | 9
    Missing | 4 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free Survival was defined as the time from the date of randomization until either documented disease progression or death due to any cause, whichever occurred first. Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, progressive disease (PD) was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS as assessed by Blinded Independent Central Review (BICR) per RECIST 1.1 is presented. PFS is reported based on the non-parametric Kaplan-Meier method. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 39 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 296 | 295
Months | 8.3 [6.7 to 9.7] | 5.4 [4.1 to 5.6]
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Superiority; p = 0.0040, Log Rank — One-sided p-value based on log-rank test stratified by Eastern Cooperative Cancer Group (ECOG) at pre-randomization visit, response at randomization and baseline PD-L1 status; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.63 to 0.93] — Based on Cox regression model with Efron's method of tie handling and with treatment as a covariate stratified by ECOG at pre-randomization visit, response at randomization and baseline PD-L1 status

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival was the time from the date of randomization to death due to any cause. OS is reported based on the non-parametric Kaplan-Meier method. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 46 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 296 | 295
Months | 19.1 [15.9 to 22.2] | 18.6 [16.0 to 21.6]
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Superiority; p = 0.5481, Log Rank — One-sided p-value based on log-rank test stratified by ECOG at pre-randomization visit, response at randomization and baseline PD-L1 status; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.83 to 1.24] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study. The number of participants who reported 1 or more AEs is presented. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study. The number of participants who discontinued study intervention due to an AE is presented. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (GHS)/ Quality of Life (QoL) (Items 29 and 30) Combined Scale Score
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to the Global Health Status GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were each scored on a 7-point scale (1=Very Poor to 7=Excellent), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score was assessed using a constrained longitudinal data analysis (cLDA) model with the patient-reported outcome (PRO) score as the response variable, and treatment, time, treatment-by-time interaction, and clinical study stratification factors as covariates. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Baseline and Week 24
Population: The analysis population consists of all randomized participants who had at least one PRO assessment available and had received at least one dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 293 | 291
Score on a Scale | -1.24 [-3.68 to 1.19] | -1.62 [-4.11 to 0.88]
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.8238, t-test, 2 sided — Based on cLDA model with the PRO scores as the response variable with covariates for treatment by time interaction, stratification factors, response at randomization, and baseline PD-L1 expression as covariates; Difference in LS Means = 0.37, 95% CI 2-sided [-2.91 to 3.66] — Based on cLDA model with the PRO scores as the response variable with covariates for treatment by time interaction, stratification factors, response at randomization, and baseline PD-L1 expression as covariates

6. Secondary Outcome: Time to True Deterioration (TTD) in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (GHS)/Quality of Life (QoL) (Items 29 and 30) Scale Score
Description: TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline in GHS (EORTC QLQ-C30 Item 29) and QoL score (EORTC QLQ-C30 Item 30). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10- point negative change (decrease) from Baseline in GHS score, will be presented. A longer TTD indicates a better outcome. TTD is reported based on the non-parametric Kaplan-Meier method. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 285 | 283
Months | 29.08 [17.94 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 29.01 [12.55 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.3083, Log Rank — Two-sided p-value based on log-rank test stratified by ECOG at pre-randomization Visit, response at randomization, and baseline PD-L1 expression; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.66 to 1.14] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG at pre-randomization Visit, response at randomization, and baseline PD-L1 expression

7. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Lung Cancer Module 13 (QLQ-LC13) Cough (Item 1) Scale Score
Description: The EORTC QLQ-LC13 is a lung cancer specific supplemental questionnaire used in combination with the EORTC QLQ-C30 questionnaire. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-LC13 cough (Item 1) score is presented. Change from baseline score was assessed using a cLDA model with the PRO score as the response variable, and treatment, time, treatment-by-time interaction, and clinical study stratification factors as covariates. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 293 | 291
Score on a Scale | 2.42 [-0.93 to 5.77] | 0.74 [-2.69 to 4.17]
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.4686, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; Difference in Least Square Means = 1.68, 95% CI 2-sided [-2.87 to 6.23] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Time to True Deterioration (TTD) in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Lung Cancer Module 13 (QLQ-LC13) Cough (Item 1) Scale Score
Description: The EORTC QLQ-LC13 is a lung cancer specific supplemental questionnaire used in combination with the EORTC QLQ-C30 questionnaire. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in cough scale score. The TTD for cough (Item 1) is presented. TTD is reported based on the non-parametric Kaplan-Meier method. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 285 | 283
Months | 24.18 [15.64 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [16.56 to NA] — Median and Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.9174, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.76 to 1.35] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Lung Cancer Module 13 (QLQ-LC13) Chest Pain (Item 10) Scale Score
Description: The EORTC QLQ-LC13 is a lung cancer specific supplemental questionnaire used in combination with the EORTC QLQ-C30 questionnaire. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-LC13 chest pain (Item 10) score is presented. Change from baseline score was assessed using a cLDA model with the PRO score as the response variable, and treatment, time, treatment-by-time interaction, and clinical study stratification factors as covariates. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 293 | 291
Score on a Scale | 6.35 [3.95 to 8.76] | 2.52 [0.06 to 4.98]
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.0245, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; Difference in Least Square Means = 3.83, 95% CI 2-sided [0.50 to 7.16] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Time to True Deterioration (TTD) in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Lung Cancer Module 13 (QLQ-LC13) Chest Pain (Item 10) Scale Score
Description: The EORTC QLQ-LC13 is a lung cancer specific supplemental questionnaire used in combination with the EORTC QLQ-C30 questionnaire. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in chest pain scale score. The TTD for chest pain (Item 10) is presented. TTD is reported based on the non-parametric Kaplan-Meier method. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 285 | 283
Months | NA [NA to NA] — Median, Lower and Upper Limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median, Lower and Upper Limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.2133, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.88 to 1.75] — [estimate comment as in outcome 6, analysis 1]

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Dyspnea (Item 8) Scale Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in EORTC QLQ-C30 dyspnea (Item 8) score will be presented. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-C30 dyspnea (Item 8) score is presented. Change from baseline score was assessed using a cLDA model with the PRO score as the response variable, and treatment, time, treatment-by-time interaction, and clinical study stratification factors as covariates. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 293 | 291
Score on a Scale | -1.08 [-4.49 to 2.34] | -1.25 [-4.74 to 2.24]
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.9381, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; Hazard Ratio (HR) = 0.18, 95% CI 2-sided [-4.27 to 4.62] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Time to True Deterioration (TTD) in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Dyspnea (Item 8) Scale Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in Item 8 scale score. The TTD for dyspnea (Item 8) is presented. TTD is reported based on the non-parametric Kaplan-Meier method. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 285 | 283
Months | NA [NA to NA] — Median, Lower and Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [14.72 to NA] — Median and Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.8464, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.72 to 1.31] — [estimate comment as in outcome 6, analysis 1]

13. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Physical Functioning (Items 1 to 5) Scale Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) score is presented. Change from baseline score was assessed using a constrained longitudinal data analysis (cLDA) model with the patient-reported outcome (PRO) score as the response variable, and treatment, time, treatment-by-time interaction, and clinical study stratification factors as covariates. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on Scale
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 285 | 283
Score on Scale | -2.04 [-4.38 to 0.31] | 0.77 [-1.62 to 3.17]
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.0870, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; Difference in Least Square Means = -2.81, 95% CI 2-sided [-6.02 to 0.41] — [estimate comment as in outcome 5, analysis 1]

14. Secondary Outcome: Time to True Deterioration (TTD) in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Physical Functioning (Items 1 to 5) Scale Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in physical functioning Items 1 to 5 scale scores. The TTD for physical functioning (Item 1-5) is presented. TTD is reported based on the non-parametric Kaplan-Meier method. Per protocol this outcome measure was not planned for the Induction Phase.
Time Frame: Up to approximately 2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Olaparib (Maintenance Phase) | Pembro + Placebo (Maintenance Phase)
Number analyzed (Participants) | 285 | 283
Months | 22.80 [10.05 to NA] — Upper Limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [27.50 to NA] — Median and Upper Limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembro + Olaparib (Maintenance Phase) vs Pembro + Placebo (Maintenance Phase); Test type: Other; p = 0.0020, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [1.18 to 2.16] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 4 years
Description: Mortality includes all enrolled participants regardless of treatment status. AEs include all participants who received ≥1 dose of study drug, counted in the latest arm for which a participant received drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs.
Groups:
- Pembro + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase): Participants received Pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) on Day 1 of each 21-day cycle for 4 cycles PLUS Carboplatin Area Under Curve (AUC) 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles PLUS investigator's choice of either Paclitaxel (200 mg/m^2 Q3W on Day 1 of each 21-day cycle for 4 cycles or Nab-paclitaxel (100 mg/m^2 Q3W on Days 1, 8, 15 of each 21-day cycle for 4 cycles). Participants may then randomize to one of the blinded treatment arms.
- Pembro+Olaparib (Maintenance Phase ): This arm includes participants who randomized following completion of the induction period. After the induction period, participants received pembrolizumab IV on Day 1 of each 21-day for up to 31 cycles PLUS maintenance oral olaparib 300 mg twice daily. In the Maintenance Phase, the participant continued to receive maintenance olaparib until centrally verified progressive disease, physician decision or intolerable toxicity.
  Participants treated with pembrolizumab who completed 35 cycles of pembrolizumab during the study with stable disease (SD), complete response (CR), or partial response (PR), and without a current adverse event (AE), may have been eligible for retreatment with up to an additional 17 cycles (approximately 1 year) of pembrolizumab if they experienced radiographic disease progression after stopping treatment in the Maintenance Phase.
- Pembro+Placebo (Maintenance Phase): This arm includes participants who randomized following completion of the induction period. After the induction period, participants received pembrolizumab IV on Day 1 of each 21-day for up to 31 cycles PLUS matching maintenance olaparib placebo twice daily. In the Maintenance Phase, the participant continued to receive maintenance olaparib placebo until centrally verified progressive disease, physician decision or intolerable toxicity.
  Participants treated with pembrolizumab who completed 35 cycles of pembrolizumab during the study with SD, CR, or PR, and without a current AE, may have been eligible for retreatment with up to an additional 17 cycles (approximately 1 year) of pembrolizumab if they experienced radiographic disease progression after stopping treatment in the Maintenance Phase.
- Pembro + Olaparib (Second Course Pembro Only); Pembro + Placebo (Second Course Pembro Only): Eligible participants who received 35 cycles of Pembrolizumab and progressed with SD, PR, or CR in either arm were eligible for an optional 1 additional year (17 cycles) of Pembrolizumab.
Arm/Group | Pembro + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase) | Pembro+Olaparib (Maintenance Phase ) | Pembro+Placebo (Maintenance Phase) | Pembro + Olaparib (Second Course Pembro Only) | Pembro + Placebo (Second Course Pembro Only)
All-Cause Mortality (participants affected / at risk) | 101/851 | 188/296 | 189/295 | 0/7 | 2/9
Serious Adverse Events (participants affected / at risk) | 220/851 | 97/294 | 77/292 | 2/7 | 1/9
Other Adverse Events (participants affected / at risk) | 787/851 | 265/294 | 240/292 | 4/7 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase) (N=851) | Pembro+Olaparib (Maintenance Phase ) (N=294) | Pembro+Placebo (Maintenance Phase) (N=292) | Pembro + Olaparib (Second Course Pembro Only) (N=7) | Pembro + Placebo (Second Course Pembro Only) (N=9)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 10 (10) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (14) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 11 (11) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 9 (9) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 10 (10) | 8 (8) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 36 (41) | 13 (14) | 11 (12) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 3 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis noninfective (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Carboplatin + Paclitaxel or Nab-Paclitaxel (Induction Phase) (N=851) | Pembro+Olaparib (Maintenance Phase ) (N=294) | Pembro+Placebo (Maintenance Phase) (N=292) | Pembro + Olaparib (Second Course Pembro Only) (N=7) | Pembro + Placebo (Second Course Pembro Only) (N=9)
Anaemia (Blood and lymphatic system disorders) | 369 (432) | 130 (215) | 45 (69) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 168 (299) | 44 (115) | 13 (19) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 23 (28) | 21 (39) | 11 (13) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 279 (520) | 57 (118) | 16 (25) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 200 (314) | 56 (127) | 19 (43) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 25 (25) | 23 (24) | 34 (38) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 147 (165) | 26 (30) | 29 (30) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 112 (148) | 23 (32) | 33 (49) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 215 (346) | 69 (98) | 35 (51) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 66 (75) | 26 (34) | 11 (15) | 0 (0) | 0 (0)
Asthenia (General disorders) | 115 (138) | 42 (50) | 37 (47) | 0 (0) | 0 (0)
Fatigue (General disorders) | 105 (136) | 32 (36) | 40 (44) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 74 (83) | 18 (21) | 16 (20) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 13 (13) | 19 (20) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 23 (26) | 17 (19) | 11 (21) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 54 (59) | 25 (32) | 29 (50) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 39 (45) | 25 (27) | 27 (42) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 38 (40) | 21 (31) | 22 (33) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 31 (37) | 26 (41) | 17 (39) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 36 (37) | 14 (14) | 15 (16) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 140 (166) | 54 (62) | 47 (53) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 33 (35) | 24 (51) | 21 (37) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 31 (34) | 15 (24) | 22 (40) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 41 (50) | 5 (5) | 18 (29) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 65 (102) | 29 (35) | 32 (47) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 20 (24) | 21 (23) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 75 (114) | 9 (10) | 16 (18) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 25 (26) | 17 (21) | 11 (11) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 19 (20) | 20 (27) | 21 (26) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (35) | 36 (46) | 37 (40) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 (38) | 29 (33) | 32 (35) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 10 (10) | 17 (23) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 55 (59) | 22 (30) | 27 (30) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 63 (66) | 22 (23) | 24 (31) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 18 (18) | 8 (8) | 7 (8) | 1 (1) | 0 (0)
Malaise (General disorders) | 27 (35) | 4 (4) | 2 (3) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 10 (11) | 4 (4) | 4 (6) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 4 (4) | 4 (4) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (10) | 9 (11) | 7 (9) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 15 (19) | 10 (11) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 8 (8) | 8 (8) | 9 (14) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8) | 6 (8) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 120 (130) | 7 (7) | 6 (7) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 60 (65) | 5 (7) | 6 (6) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 62 (65) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 43 (44) | 10 (14) | 8 (9) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 5 (6) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 279 (279) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity was not directed by the Sponsor, the investigator agreed to submit all manuscripts or abstracts to the Sponsor before submission. This allowed the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT03976362/Prot_SAP_001.pdf